CLINICAL TRIAL: NCT02814851
Title: Evaluation of Cardiac Hemodynamic Modifications During Temporary Left Atrial Appendage Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Pierre Wauthy, Head of clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUB-LAA-Ligature
Record Dates: First submitted 2016-04-20; First posted 2016-06-28 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Cardiac Surgery
Keywords: Left atrium appendage (LAA) occlusion; Transesophageal echocardiography; Cardiac output hemodynamic measurement; Leycom Pressure/Volume Combination Catheter
MeSH Terms: conditions — Bites and Stings | interventions — Echocardiography, Transesophageal; Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non valvular cardiac surgery (Experimental): The study will be conducted at the CHU Brugmann Hospital, with collaboration between cardiac surgery and cardiology wards. Subjects referred for non valvular cardiac surgery will be prospectively included during the first 6 months following the onset of the protocol.
  Interventions: Device: Transesophageal echocardiogram; Device: Thermistor-tipped catheter; Device: Pressure/volume catheter; Device: Transthoracic echocardiography

INTERVENTIONS:
Device: Transesophageal echocardiogram — All patients will undergo a standard surgical procedure by the surgical team of CHU Brugmann. A transesophageal echocardiogram (TEE) will be performed and the TEE probe will stay continuously during the entire procedure, to allow all necessary measurements.
Device: Thermistor-tipped catheter — All patients will undergo a standard surgical procedure by the surgical team of CHU Brugmann.During the procedure, a thermistor-tipped catheter (model 93A-131-7F, Edwards, Santa Ana, CA) will be inserted into the pulmonary artery to measure right atrial pressure (Pra), pulmonary arterial pressure (Ppa), Ppao and thermodilution cardiac output. Ringer's lactate will be infused to maintain an occluded pulmonary arterial pressure (Ppao) of 8-10 mmHg.
Device: Pressure/volume catheter — All patients will undergo a standard surgical procedure by the surgical team of CHU Brugmann.During the procedure, a pressure/volume catheter (CD Leicom, Zoetermeer, Netherland) will be placed in the left ventricle through a left superior pulmonary vein purse string, in order to measure alternatively LV pressure/volume loops and LA pressure.
Device: Transthoracic echocardiography — A complete transthoracic echocardiography will be performed the day before the surgical procedure. It will establish the presence of the inclusion and exclusion criteria, as stipulated above. This will be done using a Philips IE33 echocardiograph (Koninklijke Philips Electronics N.V., Netherlands).
  During the surgical procedure, a transesophageal echocardiogram will be performed, using an Acuson Sequoia system (Siemens AG, Germany).

SUMMARY:
The left atrium appendage (LAA) is a remnant of the original embryonic left atrium formed during the third week of gestation. LAA is believed to function as a decompression chamber during left ventricular systole and other periods when left atrial pressure is elevated. The LAA is also a major endocrine organ and is the main producer of ANP (atrial natriuretic peptide) in the human heart. The ANP concentration is 40 times higher in the LAA walls than in the rest of the atrial wall. A study of patients having undergone the maze procedure and associated LAA removal found a significantly lower ANP secretion and an increase in salt and water retention. Whether this could eventually lead to hypertension or heart failure symptoms is not known.

Removal of the LAA is routinely performed during antiarrhythmic surgical techniques ("MAZE surgery") to reduce the risk of subsequent LAA thrombus. Furthermore, new percutaneous ablation techniques target LAA to reduce further risks of atrial fibrilation recurrences. However, in addition to effects on diastolic atrial function and atrial natriuretic peptide (ANP) secretion, this could potentially reduce stroke volume and cardiac output and may thus promote heart failure. Its removal could be particularly detrimental in patients with existing heart failure and high intraatrial pressure, as it would further promote pulmonary congestion and also reduce their cardiac output.

The study will be conducted at the CHU Brugmann Hospital, with collaboration between cardiac surgery and cardiology wards. Subjects referred for non valvular cardiac surgery will be prospectively included during the first 6 months following the onset of the protocol. Echocardiographic and invasive data will be collected simultaneously.

The goals of the study are:

* To evaluate the immediate impact of temporary closure of the LAA using a vascular clamp in the beating heart of human subjects during cardiac surgery. Impact of LAA occlusion will be measured using transesophageal echocardiography and hemodynamic measurement of the cardiac output.
* To correlate echocardiographic parameters with in situ hemodynamic data.

A significant role of the LAA in the cardiac hemodynamic including the left ventricle outflow might have different clinical implications and will raise questions about:

* Appropriateness of LAA resection in antiarrhythmic surgery
* Importance of restoring sinus rhythm in atrial fibrilation patients
* Importance to spare LAA from ablation during atrial fibrilation ablation to avoid significant consequences on cardiac function.
* Appropriateness of the LAA occluding device in atrial fibrillation patients.

ELIGIBILITY:
Inclusion Criteria:

* Aortic valve stenosis suitable to surgery
* Left Atrium<50 mm in the parasternal long axis view
* Sinus rhythm at the time of patient's inclusion and during the procedure

Exclusion Criteria:

* Hypertrophic cardiomyopathy (diastolic septal thickness > 15mm).
* Heart failure with Left Ventricule Ejection Fraction < 45%.
* Significant mitral regurgitation/stenosis
* Significant aortic regurgitation
* History of atrial fibrillation
* Presence of prosthetic valves
* Complex congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
Left atrium (LA) dP/dt max | Baseline (before LAA clamping)
  Fluid-filled catheter-derived pressures will be zero-referenced at mid-chest level and processed using disposable transducers (Baxter-Bentley, Uden, the Netherlands) and a Sirecust 404 monitoring system (Siemens, Erlangen, Germany). Micromanometer-derived pressures and conductance catheter data will be processed using a Leicom INCA intracardiac monitor (CD Leycom, Zoetermeer, Netherlands). All pressures and volume signals will be digitalized at 200 Hz and stored in a PC for off-line analysis.
Left atrium dP/dt max | 5 minutes after LAA clamping
  Fluid-filled catheter-derived pressures will be zero-referenced at mid-chest level and processed using disposable transducers (Baxter-Bentley, Uden, the Netherlands) and a Sirecust 404 monitoring system (Siemens, Erlangen, Germany). Micromanometer-derived pressures and conductance catheter data will be processed using a Leicom INCA intracardiac monitor (CD Leycom, Zoetermeer, Netherlands). All pressures and volume signals will be digitalized at 200 Hz and stored in a PC for off-line analysis.
Left atrium output | Baseline (before LAA clamping)
  Fluid-filled catheter-derived pressures will be zero-referenced at mid-chest level and processed using disposable transducers (Baxter-Bentley, Uden, the Netherlands) and a Sirecust 404 monitoring system (Siemens, Erlangen, Germany). Micromanometer-derived pressures and conductance catheter data will be processed using a Leicom INCA intracardiac monitor (CD Leycom, Zoetermeer, Netherlands). All pressures and volume signals will be digitalized at 200 Hz and stored in a PC for off-line analysis. The cardiac output will be measured by thermodilution (REF-1 computer, Edwards, Irvine, CA).
Left atrium output | 5 minutes after LAA clamping
  Fluid-filled catheter-derived pressures will be zero-referenced at mid-chest level and processed using disposable transducers (Baxter-Bentley, Uden, the Netherlands) and a Sirecust 404 monitoring system (Siemens, Erlangen, Germany). Micromanometer-derived pressures and conductance catheter data will be processed using a Leicom INCA intracardiac monitor (CD Leycom, Zoetermeer, Netherlands). All pressures and volume signals will be digitalized at 200 Hz and stored in a PC for off-line analysis. The cardiac output will be measured by thermodilution (REF-1 computer, Edwards, Irvine, CA).
Left atrium contractility index (dP/dt max)/P | Baseline (before LAA clamping)
  Fluid-filled catheter-derived pressures will be zero-referenced at mid-chest level and processed using disposable transducers (Baxter-Bentley, Uden, the Netherlands) and a Sirecust 404 monitoring system (Siemens, Erlangen, Germany). Micromanometer-derived pressures and conductance catheter data will be processed using a Leicom INCA intracardiac monitor (CD Leycom, Zoetermeer, Netherlands). All pressures and volume signals will be digitalized at 200 Hz and stored in a PC for off-line analysis.
Left atrium contractility index (dP/dt max)/P | 5 minutes after LAA clamping
  Fluid-filled catheter-derived pressures will be zero-referenced at mid-chest level and processed using disposable transducers (Baxter-Bentley, Uden, the Netherlands) and a Sirecust 404 monitoring system (Siemens, Erlangen, Germany). Micromanometer-derived pressures and conductance catheter data will be processed using a Leicom INCA intracardiac monitor (CD Leycom, Zoetermeer, Netherlands). All pressures and volume signals will be digitalized at 200 Hz and stored in a PC for off-line analysis.
Left ventricle (LV) dP/dt max | Baseline (before LAA clamping)
  Fluid-filled catheter-derived pressures will be zero-referenced at mid-chest level and processed using disposable transducers (Baxter-Bentley, Uden, the Netherlands) and a Sirecust 404 monitoring system (Siemens, Erlangen, Germany). Micromanometer-derived pressures and conductance catheter data will be processed using a Leicom INCA intracardiac monitor (CD Leycom, Zoetermeer, Netherlands). All pressures and volume signals will be digitalized at 200 Hz and stored in a PC for off-line analysis.
Left ventricle dP/dt max | 5 minutes after LAA clamping
  Fluid-filled catheter-derived pressures will be zero-referenced at mid-chest level and processed using disposable transducers (Baxter-Bentley, Uden, the Netherlands) and a Sirecust 404 monitoring system (Siemens, Erlangen, Germany). Micromanometer-derived pressures and conductance catheter data will be processed using a Leicom INCA intracardiac monitor (CD Leycom, Zoetermeer, Netherlands). All pressures and volume signals will be digitalized at 200 Hz and stored in a PC for off-line analysis.
Left ventricle output | Baseline (before LAA clamping)
  Fluid-filled catheter-derived pressures will be zero-referenced at mid-chest level and processed using disposable transducers (Baxter-Bentley, Uden, the Netherlands) and a Sirecust 404 monitoring system (Siemens, Erlangen, Germany). Micromanometer-derived pressures and conductance catheter data will be processed using a Leicom INCA intracardiac monitor (CD Leycom, Zoetermeer, Netherlands). All pressures and volume signals will be digitalized at 200 Hz and stored in a PC for off-line analysis. The cardiac output will be measured by thermodilution (REF-1 computer, Edwards, Irvine, CA).
Left ventricle output | 5 minutes after LAA clamping
  Fluid-filled catheter-derived pressures will be zero-referenced at mid-chest level and processed using disposable transducers (Baxter-Bentley, Uden, the Netherlands) and a Sirecust 404 monitoring system (Siemens, Erlangen, Germany). Micromanometer-derived pressures and conductance catheter data will be processed using a Leicom INCA intracardiac monitor (CD Leycom, Zoetermeer, Netherlands). All pressures and volume signals will be digitalized at 200 Hz and stored in a PC for off-line analysis. The cardiac output will be measured by thermodilution (REF-1 computer, Edwards, Irvine, CA).
LV contractility index (dP/dt max)/P | Baseline (before LAA clamping)
  Fluid-filled catheter-derived pressures will be zero-referenced at mid-chest level and processed using disposable transducers (Baxter-Bentley, Uden, the Netherlands) and a Sirecust 404 monitoring system (Siemens, Erlangen, Germany). Micromanometer-derived pressures and conductance catheter data will be processed using a Leicom INCA intracardiac monitor (CD Leycom, Zoetermeer, Netherlands). All pressures and volume signals will be digitalized at 200 Hz and stored in a PC for off-line analysis. LV contractility will be estimated from the slope of the end-systolic pressure-volume relation.
LV contractility index (dP/dt max)/P | 5 minutes after LAA clamping
  Fluid-filled catheter-derived pressures will be zero-referenced at mid-chest level and processed using disposable transducers (Baxter-Bentley, Uden, the Netherlands) and a Sirecust 404 monitoring system (Siemens, Erlangen, Germany). Micromanometer-derived pressures and conductance catheter data will be processed using a Leicom INCA intracardiac monitor (CD Leycom, Zoetermeer, Netherlands). All pressures and volume signals will be digitalized at 200 Hz and stored in a PC for off-line analysis. LV contractility will be estimated from the slope of the end-systolic pressure-volume relation.
Occluded pulmonary arterial pressure (Ppao) | Baseline (before LAA clamping)
  Fluid-filled catheter-derived pressures will be zero-referenced at mid-chest level and processed using disposable transducers (Baxter-Bentley, Uden, the Netherlands) and a Sirecust 404 monitoring system (Siemens, Erlangen, Germany). Micromanometer-derived pressures and conductance catheter data will be processed using a Leicom INCA intracardiac monitor (CD Leycom, Zoetermeer, Netherlands). All pressures and volume signals will be digitalized at 200 Hz and stored in a PC for off-line analysis.
Occluded pulmonary arterial pressure (Ppao) | 5 minutes after LAA clamping
  Fluid-filled catheter-derived pressures will be zero-referenced at mid-chest level and processed using disposable transducers (Baxter-Bentley, Uden, the Netherlands) and a Sirecust 404 monitoring system (Siemens, Erlangen, Germany). Micromanometer-derived pressures and conductance catheter data will be processed using a Leicom INCA intracardiac monitor (CD Leycom, Zoetermeer, Netherlands). All pressures and volume signals will be digitalized at 200 Hz and stored in a PC for off-line analysis.

SECONDARY OUTCOMES:
Area fractional shortening (AFS) of the left atrium appendage (LAA) | Baseline (before LAA clamping)
  Transesophageal echocardiography data (Acuson Sequoia system - Siemens AG, Germany). Computed with the following formula: AFS 2CME90°= (Amax-Amin)/Amax.
Area fractional shortening (AFS) of the left atrium appendage (LAA) | 5 minutes after LAA clamping
  Transesophageal echocardiography data (Acuson Sequoia system - Siemens AG, Germany). Computed with the following formula: AFS 2CME90°= (Amax-Amin)/Amax.
Ejection volume of the LAA (left atrium appendage) | Baseline (before LAA clamping)
  Transesophageal echocardiography data (Acuson Sequoia system - Siemens AG, Germany). Computed with the following formula: LAA ejection volume= 3,14*D1*D2*TVI PW LAA/4, where D1 and D2 are the diameters of the opening of the LAA at 0° and 90°
Ejection volume of the LAA (left atrium appendage) | 5 minutes after LAA clamping
  Transesophageal echocardiography data (Acuson Sequoia system - Siemens AG, Germany). Computed with the following formula: LAA ejection volume= 3,14*D1*D2*TVI PW LAA/4, where D1 and D2 are the diameters of the opening of the LAA at 0° and 90°
Stroke volume | Baseline (before LAA clamping)
  Transesophageal echocardiography data (Acuson Sequoia system - Siemens AG, Germany). Computed with the following formula: Stroke volume= 3,14D²*Aortic PW TVI /4, where D is the LVOT (left ventricular outflow tract)diameter in A3C.
Stroke volume | 5 minutes after LAA clamping
  Transesophageal echocardiography data (Acuson Sequoia system - Siemens AG, Germany). Computed with the following formula: Stroke volume= 3,14D²*Aortic PW TVI /4, where D is the LVOT (left ventricular outflow tract) diameter in A3C.
Amplitude of the emptying pulse wave of the LAA (left atrium appendage) | Baseline (before LAA clamping)
  Transesophageal echocardiography data (Acuson Sequoia system - Siemens AG, Germany). 2C ME 90° measure
Amplitude of the emptying pulse wave of the LAA (left atrium appendage) | 5 minutes after LAA clamping
  Transesophageal echocardiography data (Acuson Sequoia system - Siemens AG, Germany). 2C ME 90° measure
TVI (Aortic Time-Velocity Integral) of the emptying pulse wave of the LAA (left atrium appendage) | Baseline (before LAA clamping)
  Transgastric or deep transgastric aortic Pulse Wave Doppler. 2C ME 90° measure
TVI (Aortic Time-Velocity Integral) of the emptying pulse wave of the LAA (left atrium appendage) | 5 minutes after LAA clamping
  Transgastric or deep transgastric aortic Pulse Wave Doppler. 2C ME 90° measure
Amplitude of the mitral A wave | Baseline (before LAA clamping)
  Amplitude A wave: measured with DTI (Tissue Doppler ) 4C ME 0° lateral ring
Amplitude of the mitral A wave | 5 minutes after LAA clamping
  Amplitude A wave: measured with DTI (Tissue Doppler ) 4C ME 0° lateral ring
TVI (Aortic Time-Velocity Integral) of the left upper pulmonary vein (LUPV) | Baseline (before LAA clamping)
  Measured by aortic Pulse Wave (PW) Doppler flow
TVI (Aortic Time-Velocity Integral) of the left upper pulmonary vein (LUPV) | 5 minutes after LAA clamping
  Measured by aortic Pulse Wave (PW) Doppler flow

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Wauthy, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Pritchett AM, Jacobsen SJ, Mahoney DW, Rodeheffer RJ, Bailey KR, Redfield MM. Left atrial volume as an index of left atrial size: a population-based study. J Am Coll Cardiol. 2003 Mar 19;41(6):1036-43. doi: 10.1016/s0735-1097(02)02981-9. PMID 12651054
- [Background] Moller JE, Hillis GS, Oh JK, Seward JB, Reeder GS, Wright RS, Park SW, Bailey KR, Pellikka PA. Left atrial volume: a powerful predictor of survival after acute myocardial infarction. Circulation. 2003 May 6;107(17):2207-12. doi: 10.1161/01.CIR.0000066318.21784.43. Epub 2003 Apr 14. PMID 12695291
- [Background] Tsang TS, Barnes ME, Gersh BJ, Takemoto Y, Rosales AG, Bailey KR, Seward JB. Prediction of risk for first age-related cardiovascular events in an elderly population: the incremental value of echocardiography. J Am Coll Cardiol. 2003 Oct 1;42(7):1199-205. doi: 10.1016/s0735-1097(03)00943-4. PMID 14522480
- [Background] Osranek M, Fatema K, Qaddoura F, Al-Saileek A, Barnes ME, Bailey KR, Gersh BJ, Tsang TS, Zehr KJ, Seward JB. Left atrial volume predicts the risk of atrial fibrillation after cardiac surgery: a prospective study. J Am Coll Cardiol. 2006 Aug 15;48(4):779-86. doi: 10.1016/j.jacc.2006.03.054. Epub 2006 Jul 25. PMID 16904549
- [Background] Tsang TS, Barnes ME, Gersh BJ, Bailey KR, Seward JB. Left atrial volume as a morphophysiologic expression of left ventricular diastolic dysfunction and relation to cardiovascular risk burden. Am J Cardiol. 2002 Dec 15;90(12):1284-9. doi: 10.1016/s0002-9149(02)02864-3. PMID 12480035
- [Background] Stollberger C, Schneider B, Finsterer J. Elimination of the left atrial appendage to prevent stroke or embolism? Anatomic, physiologic, and pathophysiologic considerations. Chest. 2003 Dec;124(6):2356-62. doi: 10.1378/chest.124.6.2356. PMID 14665520
- [Background] Al-Saady NM, Obel OA, Camm AJ. Left atrial appendage: structure, function, and role in thromboembolism. Heart. 1999 Nov;82(5):547-54. doi: 10.1136/hrt.82.5.547. PMID 10525506
- [Background] Sievert H, Lesh MD, Trepels T, Omran H, Bartorelli A, Della Bella P, Nakai T, Reisman M, DiMario C, Block P, Kramer P, Fleschenberg D, Krumsdorf U, Scherer D. Percutaneous left atrial appendage transcatheter occlusion to prevent stroke in high-risk patients with atrial fibrillation: early clinical experience. Circulation. 2002 Apr 23;105(16):1887-9. doi: 10.1161/01.cir.0000015698.54752.6d. PMID 11997272
- [Background] Akosah KO, Funai JT, Porter TR, Jesse RL, Mohanty PK. Left atrial appendage contractile function in atrial fibrillation. Influence of heart rate and cardioversion to sinus rhythm. Chest. 1995 Mar;107(3):690-6. doi: 10.1378/chest.107.3.690. PMID 7874938
- [Background] Kamohara K, Popovic ZB, Daimon M, Martin M, Ootaki Y, Akiyama M, Zahr F, Cingoz F, Ootaki C, Kopcak MW Jr, Dessoffy R, Liu J, Thomas JD, Gillinov AM, Fukamachi K. Impact of left atrial appendage exclusion on left atrial function. J Thorac Cardiovasc Surg. 2007 Jan;133(1):174-81. doi: 10.1016/j.jtcvs.2006.08.057. PMID 17198808
- [Background] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise JS, Solomon SD, Spencer KT, Sutton MS, Stewart WJ; Chamber Quantification Writing Group; American Society of Echocardiography's Guidelines and Standards Committee; European Association of Echocardiography. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. J Am Soc Echocardiogr. 2005 Dec;18(12):1440-63. doi: 10.1016/j.echo.2005.10.005. No abstract available. PMID 16376782